CLINICAL TRIAL: NCT01478412
Title: A Prospective Evaluation of Polymer Based Fiducials for Use in Imaging Patients Receiving Treatment for Prostate Cancer
Brief Title: An Evaluation of Polymer Based Fiducials for Use in Imaging Patients Receiving Treatment for Prostate Cancer
Acronym: Clarity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Chang, MD (Other)
Responsible Party: Sponsor-Investigator, John Chang, MD, John Chang, MD, ProCure Proton Therapy Center
Organization: ProCure Proton Therapy Center (Other)
Other Study IDs: CHI-001
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate cancer; Low risk; Intermediate risk; T1; T2a; T2b; Gleason 6; Gleason 7; PSA 10; PSA 20
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Males with prostate adenocarcinoma: English speaking males with histologically confirmed prostate adenocarcinoma and diagnosis of low risk or intermediate risk prostate cancer.
  Interventions: Other: Polymer based fiducial placement

INTERVENTIONS:
Other: Polymer based fiducial placement — Fiducial marker placement with rectal ultrasound imaging.

SUMMARY:
This trial is to determine if prostate target delineation obtained through an ultrasound based system is equivalent in accuracy to the MRI image fusion, and if alignment correction vectors obtained from ultrasound imaging are of equivalent accuracy to orthogonal X-ray imaging for daily prostate positioning.

DETAILED DESCRIPTION:
The investigators will also be assessing the following:

1. Whether polymer-based markers can be adequately visualized on daily stereoscopic imaging compared to gold seed markers.
2. Whether polymer-based markers are visible on ultrasound imaging.
3. To determine if the polymer-based marker produces fewer artifacts on treatment planning CT scans than gold markers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* diagnosis of low risk or intermediate risk prostate cancer
* approved for proton therapy treatment at CDH ProCure Proton Therapy Center
* prescribed and consented for the placement of fiducial markers into the prostate as part of the standard treatment procedure
* capable of receiving an MRI of the pelvis region for prostate localization
* the prostate gland of eligible patients must be capable of imaging from an anterior trans-abdominal ultrasound as determined by the treating investigator
* must be fluent in the English language; must be able to provide written study consent

Exclusion Criteria:

* Evidence of a large TURP defect per investigator discretion
* previous prostate cancer surgery including prostatectomy, hyperthermia and cryosurgery
* previous pelvic radiation for prostate cancer
* current grade 2 or above incontinence
* history of orthopedic procedures in the area of the treatment, specifically no prior hip replacement or procedure in which metallic or high density material remains which would be within stereoscopic kilovoltage imaging area
* prior permanent placement of any metallic or high density material within the prostate
* known allergy to ultrasonic gel

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of all races and ethnic groups are eligible for this trial. Since this is a prostate study, only males will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-12

PRIMARY OUTCOMES:
Ultrasound versus MRI image fusion for daily prostate positioning | 4 months
  Determine if prostate target delineation obtained through an ultrasound based system is equivalent in accuracy to the MRI image fusion method, and if alighment crrection vectors obtained from ultransound imaging are of equivalent accuracy to orthogonal X-ray imaging for daily prostate positioning.

SECONDARY OUTCOMES:
Polymer based marker visualization | 4 months
  To determine if polymer based markers can be adequately visualized on daily stereoscopic imaging compared to gold seed markers

CONTACTS AND LOCATIONS:
Overall Officials: John Chang, MD, Principal Investigator — ProCure Proton Therapy Center
Locations (1):
- ProCure Proton Therapy Center, Warrenville, Illinois, United States

REFERENCES:
- See also: ProCure Proton Therapy Center — http://www.procure.com/OurLocations/Illinois.aspx